CLINICAL TRIAL: NCT05360992
Title: Pulmonary Embolism: Mechanism and Therapeutic Innovation
Status: Completed | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Lu Hua, Director, Center for Respiratory and Pulmonary Vascular Diseases，Principal Investigator, Clinical Professor, China National Center for Cardiovascular Diseases
Other Study IDs: 2017-I2M-3-003
Record Dates: First submitted 2022-04-27; First posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Pulmonary Embolism
Keywords: pulmonary embolism; chronic thromboembolic pulmonary hypertension; mechanism; therapy; outcome
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — storage at -80℃
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To explore the pathogenesis, therapy and outcome of pulmonary embolism (PE) and chronic thromboembolic pulmonary hypertension (CTEPH).

DETAILED DESCRIPTION:
The study recruited consecutive outpatients or hospitalized patients diagnosed with pulmonary embolism (PE cohort) and chronic thromboembolic pulmonary hypertension (CTEPH cohort). The follow-up of all patients was performed annually by phone or outpatient visit. The main outcomes were bleeding, recurrent events, and survival. The objective of the study was to explore the pathogenesis, therapy and outcome of PE and CTEPH.

ELIGIBILITY:
Inclusion Criteria:

* All hospitalized patients or outpatients diagnosed with PE or CTEPH;
* Age ≥18.

Exclusion Criteria:

* Refused informed consents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The consecutive hospitalized patients or outpatients diagnosed with PE or CTEPH.
Sampling Method: Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2021-10-13 (Actual)

PRIMARY OUTCOMES:
Recurrent Incidence of Patients | through study completion, an average of 1 year.
  Recurrent PE was measured by computed tomography pulmonary angiography (CTPA) or ventilation/perfusion (V/Q) lung scans. Recurrent deep venous thrombosis was measured by lower extremity Doppler ultrasound.
Bleeding Rate of Patients | through study completion, an average of 1 year.
  Events were recored by follow-up.
Survival Rate of Patients | through study completion, an average of 1 year.
  Events were recored by follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Lu Hua, Dr., Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital

REFERENCES:
- [Derived] Wu Y, Hu S, Yan XX, Peng FH, Tan JS, Guo TT, Gao X, Hua L. Chronic Thromboembolic Pulmonary Hypertension in Females: Clinical Features and Survival. J Cardiovasc Dev Dis. 2022 Sep 16;9(9):308. doi: 10.3390/jcdd9090308. PMID 36135453